CLINICAL TRIAL: NCT05533073
Title: Comparative Bioavailability Study Between Etoricoxib 90 mg and Tramadol 50 mg, Administered Individually or in Combination, Single Dose in Healthy Subjects of Both Genders Under Fasting Conditions
Brief Title: Comparative Bioavailability Study Between Etoricoxib and Tramadol, Administered Individually or in Combination
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BD ET-Sil No. 112-19
Record Dates: First submitted 2022-09-06; First posted 2022-09-08 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Healthy
Keywords: Pharmacokinetic; Bioavailability; Fixed-dose combination (FDC); Etoricoxib; Tramadol; Pain
MeSH Terms: conditions — Pain | interventions — Tramadol; Etoricoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Etoricoxib/Tramadol FDC (Experimental): Pharmaceutical Form: Sachet with granules to dilute in 100 mL of water Formula: Each sachet contains Etoricoxib 90 mg / Tramadol 50 mg Dosage: 100 mL Administration way: oral
  Interventions: Drug: A1: Etoricoxib / Tramadol Fixed dose combination
- Group B: Etoricoxib (Active Comparator): Pharmaceutical Form: Tablet Formula: Tablet containing Etoricoxib 90 mg Dosage: 1 tablet of 90 mg Administration way: oral
  Interventions: Drug: A2: Etoricoxib
- Group C: Tramadol (Active Comparator): Pharmaceutical Form: Capsule Formula: Each capsule contains 50mg of Tramadol Dosage:1 capsule of 50 mg Administration way: oral
  Interventions: Drug: A3: Tramadol

INTERVENTIONS:
Drug: A1: Etoricoxib / Tramadol Fixed dose combination — Sachet with granules (Laboratorios Silanes S.A. de C.V.). Formula : 90 mg/ 50 mg Pharmaceutical Form: Sachet with granules Dosage: 100 mL (90 mg/ 50mg) Administration way: oral
  Other Names: E/T
  Arms: Group A: Etoricoxib/Tramadol FDC
Drug: A2: Etoricoxib — Arcoxia®, Schering Plough S.A. de C.V. A2: Pharmaceutical Form: Tablet Formula: 90 mg Dosage: 1 tablet of 90 mg Administration way: oral
  Other Names: Arcoxia®
  Arms: Group B: Etoricoxib
Drug: A3: Tramadol — Tradol®, from Grünenthal GMBH. Pharmaceutical Form: Capsule Formula: Each capsule contains 50 mg Dosage: 1 capsule of 50 mg Administration way: oral
  Other Names: Tradol®
  Arms: Group C: Tramadol

SUMMARY:
Study carried out in the Clinical and Analytical Unit of the Department of Pharmacology and Toxicology of the Faculty of Medicine of the Autonomous University of Nuevo León, with the objective of comparing the bioavailability (Cmax, AUC) of an oral formulation containing Etoricoxib 90 mg / Tramadol 50 mg in combination with that of two oral formulations, Etoricoxib 90 mg or Tramadol 50 mg, administered as a single dose, in healthy subjects under fasting conditions.

DETAILED DESCRIPTION:
The study design was a crossover, 3 x 6 x 3, open-label, prospective and longitudinal, truncated, single-dose combination of Etoricoxib 90 mg / Tramadol 50 mg administered orally versus each component administered individually, with three treatments, three periods. , six sequences with an elimination period (washout) of 14 days and with a total of 42 healthy subjects, of both genders, under fasting conditions. Among the objectives were the characterization of the pharmacokinetic parameters, Cmax, AUC 0-72, Tmax, Ke and T1/2 of Etoricoxib and Tramadol after oral administration in a single dose, in combination: sachet with granules equivalent to Etoricoxib 90 mg/ Tramadol 50 mg manufactured by Laboratorios Silanes, S.A. of C.V. versus each component administered individually: Etoricoxib 90 mg tablet (Arcoxia®) manufactured by Schering Plough S.A de C.V. and Tramadol 50 mg capsule (Tradol®) made by Grunenthal GMBH (private company).

ELIGIBILITY:
Inclusion Criteria:

* The subjects must have been accepted by the COFEPRIS (Federal Commission for the Protection against Sanitary Risks) research subjects registration database.
* Subjects without a subordinate relationship with the researchers.
* Subjects who have given informed consent in writing.
* Subjects of both genders, aged between 18 and 55 years, Mexicans. - -Subjects with no background of hypersensitivity or allergies to the drug under study or related drugs.
* Body mass index between 18 and 27 kg/m2.
* Healthy subjects, according to the results of the complete clinical history, electrocardiogram and the integration of the results of the clinical analyses, carried out in certified clinical laboratories, without alterations that require a medical intervention as a consequence.
* Subjects with negative results for immunological tests (Anti-HIV, Anti-hepatitis B and C, VDRL).
* Subjects with negative results in drug abuse screening tests: tetrahydrocannabinoids, cocaine and amphetamines.
* Negative (qualitative) pregnancy test for women of childbearing potential without Bilateral tubal obstruction or hysterectomy.
* In the case of women of childbearing age, they must have a birth control method, including barrier methods, non-hormonal intrauterine device, or bilateral tubal obstruction.

Exclusion Criteria:

* Subjects with recent history or physical examination evidence of gastrointestinal, renal, hepatic, endocrine, respiratory, cardiovascular, dermatological, or hematological disease that could affect the pharmacokinetic study of the product in research.
* Subjects who have been exposed to drugs known as liver enzyme inducers or inhibitors or who have taken drugs potentially toxic within 30 days before the start of the study.
* Subjects who have received any medication during the 7 days before the start of the study.
* Subjects who have been hospitalized for any problem during the three months before the start of the study.
* Subjects who have been rejected by the registry database of research subjects of COFEPRIS, for having participated in a clinical study within the three months prior to the start of the study.
* Subjects who have received investigational drugs within the previous 60 days th the start of the study.
* Subjects allergic to the study drug or related drugs.
* Subjects who have ingested alcohol or drinks containing xanthines (coffee, tea, cocoa, chocolate, cola) or who have eaten charcoal-grilled food or grapefruit juice , at least 10 hours before the start of the study or who have smoked tobacco 24 hours before to the start of the internment period.
* Subjects who have donated or lost 450 mL or more of blood within the previous 60 days of the beginning of the study.
* Subjects with a history of drug and/or alcohol abuse according to the DSM-IV-TR (Diagnostic and Statistical Manual of Mental Disorders) Criteria.
* Research subjects who presents alterations in the vital signs recorded during the selection.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2020-09-07 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Maximum observed concentration following the treatment (Cmax) | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose Etoricoxib/Tramadol, employing the maximum observed concentration following the treatment (Cmax), obtained graphically, from the plasma concentration profile with respect to time.
The area under the curve from time zero to the last measurable concentration (AUC 0-t) | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Etoricoxib/Tramadol, employing the area under the curve from time zero to the last measurable concentration (AUC 0-t) using the linear trapezoidal method.
The area under the curve from time zero to infinity calculated (AUC 0-inf), | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Etoricoxib/Tramadol, employing the area under the curve from time zero to infinity calculated (AUC 0-inf).
Time of the maximum measured concentration (Tmax). | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Etoricoxib/Tramadol, employing time of the maximum measured concentration (tmax), Obtained graphically, from the plasma concentration profile with respect to time.
Elimination rate (Ke) | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the fixed dose pharmacokinetics profile of Etoricoxib/Tramadol, employing the elimination rate (Ke), estimated from the terminal linear portion of the plasma concentration profile with respect to time (on a semi-log scale)
Half time elimination (t1/2) | Baseline, 0.25, 0.50, 0.75, 1.00, 1.50, 2.0, 2.5, 3.0, 4.0, 6.0, 8.0, 12,0, 15.0, 24.0, 30.0, 36.0, 48.0 and 72.0 hours.
  Evaluate the pharmacokinetics profile of the fixed dose Etoricoxib/Tramadol, employing the half time elimination (t1/2) by the quotient of Ln(2)Ke.

SECONDARY OUTCOMES:
Determine the frequency of occurrence of adverse events | 1, 15 and 29 days
  The percentage of frequency of appearance of each adverse event was evaluated.
Adverse Events | 1, 15 and 29 days
  Any adverse event were classified by severity, treatment and its relationship with the study drug was evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes Garza Ocaña, M.D, Principal Investigator — Department of Pharmacology and Toxicology of the Faculty of Medicine of the U.A.N.L
Locations (1):
- Laboratorio Silanes, S.A. de C.V., Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenthal R. An application of the Kolmogorov-Smirnov test for normality with estimated mean and variance. Psychol Rep. 1968 Apr;22(2):570. doi: 10.2466/pr0.1968.22.2.570. No abstract available. PMID 5650254
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Hauck WW, Anderson S. A new statistical procedure for testing equivalence in two-group comparative bioavailability trials. J Pharmacokinet Biopharm. 1984 Feb;12(1):83-91. doi: 10.1007/BF01063612. PMID 6747820
- [Background] Shohag MH, Islam MS, Ahmed MU, Joti JJ, Islam MS, Hasanuzzaman M, Hasnat A. Pharmacokinetic and bioequivalence study of etoricoxib tablet in healthy Bangladeshi volunteers. Arzneimittelforschung. 2011;61(11):617-21. doi: 10.1055/s-0031-1300564. PMID 22232850
- [Background] Agrawal NG, Porras AG, Matthews CZ, Rose MJ, Woolf EJ, Musser BJ, Dynder AL, Mazina KE, Lasseter KC, Hunt TL, Schwartz JI, McCrea JB, Gottesdiener KM. Single- and multiple-dose pharmacokinetics of etoricoxib, a selective inhibitor of cyclooxygenase-2, in man. J Clin Pharmacol. 2003 Mar;43(3):268-76. doi: 10.1177/0091270003251122. PMID 12638395
- [Background] Silva Mde F, Schramm SG, Kano EK, Mori Koono EE, Porta V, dos Reis Serra CH. Bioequivalence evaluation of single doses of two tramadol formulations: a randomized, open-label, two-period crossover study in healthy Brazilian volunteers. Clin Ther. 2010 Apr;32(4):758-65. doi: 10.1016/j.clinthera.2010.03.016. PMID 20435245